CLINICAL TRIAL: NCT02985489
Title: Preoperative PN Therapy in Malnourished Patients With IBD - A Randomized Controlled Trial
Brief Title: Pre-Operative Parenteral Nutrition in Malnourished Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruited
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB16-2059
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition; Inflammatory Bowel Disease 1
MeSH Terms: conditions — Malnutrition; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Participants assigned to the experimental group will commence Olimel Parenteral Nutrition therapy delivered through central venous catheter (CVC) access within 24-48 hours of admission.
  Interventions: Dietary Supplement: Olimel Parenteral Nutrition
- Control Group (No Intervention): Participants assigned to the control group will receive standard of care (SOC) nutritional therapy. Control group patients will be assessed by the RD assigned to the medical unit to which the patient has been admitted (independent RD assessment). The unit RD will follow standard nutrition screening processes to determine nutrition risk, followed by a complete nutrition assessment in the presence of nutrition risk.

INTERVENTIONS:
Dietary Supplement: Olimel Parenteral Nutrition — Olimel 5.7% with electrolytes
  Arms: Experimental Group

SUMMARY:
Malnourished patients with IBD that receive pre-operative parenteral nutrition therapy will have fewer post-operative complications compared to malnourished patients that receive standard of care nutritional therapy.

DETAILED DESCRIPTION:
Primary Objective To determine the impact of pre-operative PN therapy in malnourished patients with IBD compared with standard of care nutritional therapy on the development of total post-operative complications.

Secondary Objectives To assess the impact of pre-operative PN therapy in malnourished patients with IBD compared with standard of care nutritional therapy on the incidence of post-operative infectious complications Primary Endpoint The primary endpoints will be the incidence of post-surgical complications in malnourished patients receiving pre-operative PN therapy compared with standard of care therapy Secondary Endpoints The secondary endpoints will be the cumulative incidence of post-operative infectious complications in IBD patients receiving surgery and hospital length of stay in patients receiving pre-operative PN therapy compared to standard of care nutritional therapy METHODS Study Design This is a prospective multi-center randomized controlled study. Allocation to either intervention or control group will be randomized based on blocks system (size of 4). The randomization sequence will be computer generated. Conjoint Ethics Review Board Approval for the study protocol will be sought in conventional manner.

Withdrawal Criteria

(a) If there is any catheter - related complications (including infection) resulting in catheter removal; (b) If the patient does not meet the goal therapeutic PN rate; (c) If the duration between the PN initiation and the surgery is less than 7 days (e.g. if the patient needed an emergency surgical intervention)

Recruitment and Consent The overwhelming majority of patients with IBD are admitted to the Gastroenterology Inpatient Service. As such, recruitment to this study will take a multi-pronged approach and be stream-lined. All Gastroenterologists and Gastroenterology (GI) Fellows in training at the FMC and PLC will be made aware of the protocol and as they are rounding, they will be aware to ask any eligible patients if they would be willing to speak with our research assistant about study participation. In addition, the research coordinator assigned to the study will review the inpatient electronic medical record, Sunrise Clinical Manager (SCM) daily to identify newly admitted inpatients to both study sites with IBD. The research coordinator will review the study eligibility of the newly admitted inpatients with the GI Fellows rotating on the GI service, and approach patients for protocol review and consent once deemed eligible. All participants will undergo prospective consenting via a written informed consent either by themselves or their family members.

Study Intervention Experimental Group Participants assigned to the experimental group will commence PN therapy delivered through central venous catheter (CVC) access within 24-48 hours of admission. For the study, Olimel will be used as the PN formulation of choice. Specifically, Olimel 5.7% with electrolytes will be the preferred study product. CVC access is readily obtained at the FMC and PLC within this duration through a central venous access team designated team for this purpose. A registered dietitian (RD) will be specifically recruited for this study and will prescribe PN for eligible patients based on individualized nutritional assessment. Eligible patients will be malnourished by definition, resulting in conservative initial PN dosing to minimize the risk of refeeding syndrome . The study RD will calculate energy requirements based on predictive equations, such as the Harris Benedict Equation to determine target goals. The target protein and calorie requirements will be met within 48-72 hours of PN initiation. The optimal duration of delivery of PN preoperatively was defined by Klein et al , supported by an earlier meta-analysis by Detsky et al. The Klein meta-analysis of 14 prospective randomized trials showed a consistent benefit from preoperative PN, showing a 10% reduction in overall postoperative complications. Thirteen of 14 studies in this meta-analysis provided PN for at least 7 days , leading the Klein suggestions that use of PN should not be considered unless the duration of therapy was anticipated to be a minimum of 7 days. In accordance, PN will be administered for a minimum of 7-days prior to surgery.

Control Group Participants assigned to the control group will receive standard of care (SOC) nutritional therapy. Control group patients will be assessed by the RD assigned to the medical unit to which the patient has been admitted (independent RD assessment). The unit RD will follow standard nutrition screening processes to determine nutrition risk, followed by a complete nutrition assessment in the presence of nutrition risk. Conventionally, patients will complete calorie counts with clinical observation by the unit RD, with nutrition support, typically enteral nutrition recommended when oral intake is inadequate. Failure of EN to meet goal calorie intake may result in PN therapy at the discretion of the unit RD and treating team.

ELIGIBILITY:
Inclusion Criteria:

* (a) Age > 18 years;
* (b) Ability to provide informed consent;
* (c) Documented diagnosis of IBD as confirmed in the patient chart;
* (d) Malnourished status as defined by SGA B or C status;
* (e)Referral to colorectal surgery for surgical assessment;
* (f) No major contraindications to PN

Exclusion Criteria:

* (a) Active sepsis defined by positive blood cultures or fever > 38.5 within 48 hours of PN initiation;
* (b)Well-nourished status defined as SGA-A;
* (c) Inadequate vascular access;
* (d) Advanced liver disease;
* (e)Poorly controlled blood sugars

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of post-surgical complications in malnourished patients receiving pre-operative PN therapy compared with standard of care therapy | From date of randomization until the date of hospital discharge, assessed up to 6 months
  To determine the impact of pre-operative PN therapy in malnourished patients with IBD compared with standard of care nutritional therapy on the development of total post-operative complications.

SECONDARY OUTCOMES:
cumulative incidence of post-operative infectious complications in IBD patients receiving surgery | From date of randomization until the date of hospital discharge, assessed up to 6 months
  To assess the impact of pre-operative PN therapy in malnourished patients with IBD compared with standard of care nutritional therapy on the incidence of post-operative infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Maitreyi Raman, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No